CLINICAL TRIAL: NCT07171437
Title: Assessment of Gastrointestinal Vasculopathy in Systemic Sclerosis and Its Multisystem Correlations
Brief Title: Assessment of GIT Vasculopathy in SSc and Its Multisystem Correlations
Status: Not yet recruiting | Type: Observational
Sponsor: Esraa Moustafa Mohammed (Other)
Responsible Party: Sponsor-Investigator, Esraa Moustafa Mohammed, Specialist of Rheumatology, Assiut University
Organization: Assiut University (Other)
Other Study IDs: GIT Vasculopathy in SSc
Record Dates: First submitted 2025-09-06; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis Associated GIT Vasculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1-Study group will be undergoing to general assessment, laboratory assessment and imaging
  Interventions: Device: Doppler ultra sound
- Study group (37 patients) and control group (37 participants): Study group will be undergoing clinical assessment including
  Interventions: Device: Doppler ultra sound

INTERVENTIONS:
Device: Doppler ultra sound — - Doppler Ultrasound (DUS) To evaluate the abdominal aorta and the 3 main splanchnic vessels: Celiac Trunk (CT) Superior Mesenteric Artery (SMA) Inferior Mesenteric Artery (IMA) An ultrasound examination will be performed after a fasting period of at least 8 hours by a single operator blinded to clinical features. For abdominal vessels, the following parameters were measured: caliber, thickness, echogenicity, peak systolic velocity (PSV), end diastolic velocity (EDV), reverse velocity (RV), mean velocity (MV), resistive index (RI), and pulsatility index (PI).

SUMMARY:
* Evaluation of splanchnic vasculature, including arterial blood flow using Doppler ultrasound in patients with systemic sclerosis compared to healthy subjects.
* Correlation of Doppler findings of splanchnic vessels with GIT manifestations.
* Correlation of Doppler findings of splanchnic vessels with macrovascular affection (chest, cardiac, and renal), microvascular involvement (capillaroscopy findings), and autoantibodies (anti-SCL70 antibody and anti-centromere antibody).

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a rare, chronic autoimmune disease characterized by a complex pathophysiology involving humoral and cellular immunity, endothelial cells, and fibroblasts, leading to widespread vascular injury and excessive deposition of collagen fibers in the skin and major internal organs.

Vasculopathy is one of the main hallmarks of SSc; an early and accelerated atherosclerosis has been described in SSc; the underlying vasculopathy leads to significant impairment of blood flow due to the combined macro- and microvascular involvement. This vascular pathology may involve major organs such as the lungs, heart, GIT, and kidneys. While clinical observations and basic studies suggest that microvascular vasculopathy is of paramount importance throughout all the phases of SSc, increasing evidence suggests that macrovascular involvement also plays a critical role in the disease. Gastrointestinal (GI) involvement is highly prevalent, affecting up to 90% of SSc patients. It often remains subclinical until significant tissue damage has occurred, due to the progression of vasculopathy and fibrosis. Once symptoms develop, SSc-related GI involvement significantly worsens morbidity and mortality, patients frequently suffer marked emotional and social burdens, and advanced GI disease correlates with a more than twofold increased risk of death. The GI manifestations of SSc are heterogeneous, with possible involvement at any level, from the oral cavity down to the esophagus, stomach, small and large intestines, as well as the liver and pancreas, causing several clinical manifestations.

Upper GI involvement may result in esophageal dysmotility, gastroesophageal reflux disease (GERD), gastroparesis, GI bleeding due to esophagitis, esophageal or gastric ulcers, or gastric antral vascular ectasia (GAVE). Moreover, esophageal dysfunction has been closely linked to interstitial lung disease, indicating a possible pathogenic relationship. Lower GI-tract involvement (i.e., small intestine, large intestine, and anorectal) can also be severe, with complications including small intestinal bacterial overgrowth (SIBO), intestinal pseudo-obstruction, intestinal pneumatosis, and fecal incontinence. Impaired GI perfusion may be linked to motility disorders, which are key contributors to stasis, bowel dilation, bacterial overgrowth, malabsorption, weight loss, and ultimately reduced survival rate.

Early recognition of GI involvement is essential for symptom control and the prevention of complications. However, the diagnosis of GI involvement is challenging because it is often delayed by the lack of signs and symptoms early in the disease. Moreover, several diagnostic investigations that are useful in defining GI involvement are either invasive, expensive, or not very informative.

The involvement of the splanchnic circulation has only recently gained attention, despite vasculopathy being a systemic feature of SSc.

The vasculature of the GI tract can be evaluated noninvasively using abdominal Doppler ultrasound (DUS), a valuable tool that enables assessment of the GI vasculature and associated structures, including extra-intestinal features and splanchnic vessels. DUS measures signals from visceral vessels supplying the GI tract and evaluates the celiac trunk (CT), superior mesenteric artery (SMA), and inferior mesenteric artery (IMA) using pulsed Doppler scanning. It provides several quantifiable hemodynamic parameters, such as peak systolic, mean, and end-diastolic velocities, resistive index (RI), pulsatility index (PI), and blood flow volume.

Few studies have specifically investigated vascular abnormalities in the small and large intestines, particularly those affecting the superior and inferior mesenteric arteries. Among them, only one study has examined the correlation between DUS parameters of these mesenteric arteries and the involvement of other organs.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 years or older.
2. Patients classified as systemic sclerosis (SSc) according to ACR/EULAR 2013 classification criteria.
3. Patients who consented to undergo Doppler ultrasound (DUS) assessment of the splanchnic vessels.

Exclusion Criteria:

1. Patients younger than 18 years old.
2. Pregnancy or lactation.
3. Patients with overlapping autoimmune diseases (e.g., lupus, rheumatoid arthritis).
4. Patients with known gastrointestinal disorders not related to systemic sclerosis (e.g., inflammatory bowel disease, celiac disease).
5. Patients with a history of major gastrointestinal surgery (e.g., bowel resection).
6. Patients with diabetes mellitus (due to its independent effects on vascular flow).
7. Presence of severe comorbidities (e.g., end-stage renal disease, decompensated heart failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years or older classified as systemic sclerosis (SSc) according to ACR/EULAR 2013 classification criteria subject to in- hospital care due to SSc at Assiut University Hospital will be undergoing to clinical assessment, laboratory assessment and imaging
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of splanchnic vasculature, including arterial blood flow by Doppler ultrasound in SSc patients compared to healthy controls, and its correlation with GIT manifestations. | baseline

SECONDARY OUTCOMES:
Correlation of Doppler findings of splanchnic vessels with macrovascular affection (chest, cardiac, and renal), microvascular involvement (capillaroscopy findings), and autoantibodies (anti-SCL70 antibody and anti-centromere antibody). | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Assiut, 71111, Asyut, Egypt

REFERENCES:
- [Background] Bandini G, Monami M, Ciuti G, Mercatelli P, Lo Cricchio A, De Santis MC, Bonomi F, Bellando Randone S, Campochiaro C, El Aoufy K, Ruaro B, Giuggioli D, Hughes M, McMahan ZH, Benfaremo D, Moroncini G, Maconi G, Accogli E, Dagna L, Matucci Cerinic M, Moggi Pignone A. Doppler ultrasound, a noninvasive tool for the study of mesenteric arterial flow in systemic sclerosis: a cross-sectional study of a patient cohort with review and meta-analysis of the literature. Intern Emerg Med. 2025 Mar;20(2):381-394. doi: 10.1007/s11739-024-03783-5. Epub 2024 Oct 16. PMID 39412608
- [Background] Bandini G, Campochiaro C, Ciuti G, Baccellieri D, Ardita V, Bellando Randone S, El Aoufy K, Giuggioli D, Orlandi M, Dagna L, Chiesa R, Matucci Cerinic M, Moggi Pignone A. Doppler ultrasound unveils splanchnic arteries ischemia allowing early successful revascularization in symptomatic systemic sclerosis patients. Eur J Intern Med. 2025 May;135:126-129. doi: 10.1016/j.ejim.2025.03.019. Epub 2025 Mar 25. PMID 40140335
- [Background] McMahan Z, Pandolfino J, Perlman H, Del Galdo F, Hinchcliff M. Gastrointestinal disease in systemic sclerosis: the neglected organ system? Curr Opin Rheumatol. 2024 Nov 1;36(6):374-378. doi: 10.1097/BOR.0000000000001052. Epub 2024 Aug 28. PMID 39193877
- [Background] Keringer P, Kovacs KT, Nagy G, Agoston-Szabo A, Filipanits K, Kiss FI, Szabo A, Kumanovics G. Patient-reported gastrointestinal involvement is associated with reduced quality of life and disability in systemic sclerosis. J Scleroderma Relat Disord. 2025 Jun 5:23971983251345284. doi: 10.1177/23971983251345284. Online ahead of print. PMID 40488215